CLINICAL TRIAL: NCT04687917
Title: The Substance Abuse Treatment to HIV Care II (SAT2HIV-II) Project
Acronym: SAT2HIV-II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Alicia Bunger, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01DA052294 (NIH); R01DA052294 (NIH)
Record Dates: First submitted 2020-12-18; First posted 2020-12-29 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders | interventions — Referral and Consultation

STUDY DESIGN:
Intervention Model Description: Cluster-randomized trial
Who Masked: Outcomes Assessor
Masking Description: Single blind masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Facilitation, Training, Feedback, and Consultation (FTFC) Staff (Active Comparator): A multilevel implementation strategy
  Interventions: Behavioral: The facilitation, training, feedback, and consultation (FTFC) Strategy
- Facilitation, Training, Feedback, Consultation, and Incentivization (FTFCI) Staff (Experimental): An enhanced version of the multilevel implementation strategy
  Interventions: Behavioral: The facilitation, training, feedback, consultation, and incentivization (FTFCI) Strategy
- Facilitation, Training, Feedback, and Consultation (FTFC) Clients (Active Comparator): Clients served within the context of a multilevel implementation strategy
  Interventions: Behavioral: The facilitation, training, feedback, and consultation (FTFC) Strategy
- Facilitation, Training, Feedback, Consultation, and Incentivization (FTFCI) Clients (Experimental): Clients served within the context of an enhanced multilevel implementation strategy
  Interventions: Behavioral: The facilitation, training, feedback, consultation, and incentivization (FTFCI) Strategy

INTERVENTIONS:
Behavioral: The facilitation, training, feedback, and consultation (FTFC) Strategy — A multilevel implementation strategy that includes team-focused facilitation, as well as staff-focused training, feedback, and consultation
  Arms: Facilitation, Training, Feedback, and Consultation (FTFC) Clients; Facilitation, Training, Feedback, and Consultation (FTFC) Staff
Behavioral: The facilitation, training, feedback, consultation, and incentivization (FTFCI) Strategy — A multilevel implementation strategy that includes team-focused facilitation, as well as staff-focused training, feedback, consultation, and incentivization.
  Arms: Facilitation, Training, Feedback, Consultation, and Incentivization (FTFCI) Clients; Facilitation, Training, Feedback, Consultation, and Incentivization (FTFCI) Staff

SUMMARY:
An experiment to test the effectiveness of providing monetary bonuses to staff for achieving pre-defined performance targets regarding the implementation of a motivational interviewing-based brief intervention for substance use.

DETAILED DESCRIPTION:
A cluster-randomized type 3 hybrid trial with HIV service organizations across the United States. The primary aims is to test the effectiveness of an innovative pay-for-performance (P4P) strategy for improving the implementation of a motivational interviewing-based brief intervention for substance use.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for staff participants:

  * 18+ years of age

Inclusion criteria for client participants:

* 18+ years of age
* Diagnosed with HIV

Exclusion Criteria:

* Exclusion criteria for staff participants:

  * None

Exclusion criteria for client participants:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2026-05-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan R Garner, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
After deidentification, all of the individual participant data collected during the trial.
Time Frame: After study completion
Access Criteria: Anyone who wishes to access the data.
URL: https://www.icpsr.umich.edu/web/pages/NAHDAP/index.html

REFERENCES:
- [Derived] Garner BR, Bouris A, Charlebois ED, Li DH, Dakin A, Moskowitz J, Benbow N, Christopoulos K, Hickey MD, Imbert E. The Strategies Timeline and Activities Reporting Tables: Improving HIV Care by Improving the Reporting of Implementation Strategies. J Acquir Immune Defic Syndr. 2025 Apr 15;98(5S):e205-e215. doi: 10.1097/QAI.0000000000003613. PMID 40163072
- [Derived] Garner BR, Tueller SJ, Bradshaw M, Speck KJ, Satre D, Rash C, Donohoe T, Mungo J, Philbrick S, Ruwala R, Roosa MR, Zehner M, Ford JH 2nd. Testing the incremental effectiveness of pay-for-performance to improve implementation of a motivational interviewing brief intervention for substance use disorders in HIV settings: Results of a parallel cluster-randomized type 3 hybrid trial. Res Sq [Preprint]. 2024 Aug 9:rs.3.rs-4614222. doi: 10.21203/rs.3.rs-4614222/v1. PMID 39149465
- [Derived] Garner BR, Tueller S, Bradshaw M, Speck K, Satre D, Rash C, Donohoe T, Mungo J, Philbrick S, Ruwala R, Roosa M, Zehner M, Ford J 2nd. Testing the incremental effectiveness of pay-for-performance to improve implementation of a motivational interviewing brief intervention for substance use disorders in HIV settings: Results of a cluster-randomized type 3 hybrid trial. Res Sq [Preprint]. 2023 Dec 20:rs.3.rs-3685134. doi: 10.21203/rs.3.rs-3685134/v1. PMID 38196639

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: HIV Service Organizations (HSOs)
Groups:
- Facilitation, Training, Feedback, and Consultation (FTFC): A multilevel implementation strategy
  The facilitation, training, feedback, and consultation (FTFC) Strategy: A multilevel implementation strategy that includes team-focused facilitation, as well as staff-focused training, feedback, and consultation
- Facilitation, Training, Feedback, Consultation, and Incentivization (FTFCI): A multilevel implementation strategy
  The facilitation, training, feedback, consultation, and incentivization (FTFCI) Strategy: A multilevel implementation strategy that includes team-focused facilitation, as well as staff-focused training, feedback, consultation, and incentivization.
Period: Overall Study
Arm/Group | Facilitation, Training, Feedback, and Consultation (FTFC) | Facilitation, Training, Feedback, Consultation, and Incentivization (FTFCI)
Started | 161; 13 HIV Service Organizations (HSOs) (HIV Service Organizations (HSOs) were the unit of randomization, with both HSO staff participants and HSO client participants being cluster-randomized within each HSO.) | 267; 13 HIV Service Organizations (HSOs) (HIV Service Organizations (HSOs) were the unit of randomization, with both HSO staff participants and HSO client participants being cluster-randomized within each HSO.)
HSO Staff Participants | 44; 13 HIV Service Organizations (HSOs) | 43; 13 HIV Service Organizations (HSOs)
HSO Client Participants | 117; 13 HIV Service Organizations (HSOs) | 224; 13 HIV Service Organizations (HSOs)
Completed | 67; 13 HIV Service Organizations (HSOs) | 113; 13 HIV Service Organizations (HSOs) (This is the number of clients who consented to participate in the study, screened eligible, received the project's brief intervention, and completed the post-baseline follow-up.)
Not Completed | 94; 0 HIV Service Organizations (HSOs) | 154; 0 HIV Service Organizations (HSOs)

BASELINE CHARACTERISTICS:
Population: This study includes cluster-randomization of both staff participants and client participants. For each of the two implementation strategy conditions we have separated staff participants from client participants.
Groups:
- Facilitation, Training, Feedback, and Consultation (FTFC) Staff: A multilevel implementation strategy provided to staff
  The facilitation, training, feedback, and consultation (FTFC) Strategy: A multilevel implementation strategy that includes team-focused facilitation, as well as staff-focused training, feedback, and consultation
- Facilitation, Training, Feedback, and Consultation (FTFC) Clients: A multilevel implementation strategy that client participants are cluster-randomized
  The facilitation, training, feedback, and consultation (FTFC) Strategy: A multilevel implementation strategy that includes team-focused facilitation, as well as staff-focused training, feedback, and consultation
- Facilitation, Training, Feedback, Consultation, and Incentivization (FTFCI) Clients: An enhanced version of the multilevel implementation strategy that client participants are cluster-randomized.
  The facilitation, training, feedback, consultation, and incentivization (FTFCI) Strategy: A multilevel implementation strategy that includes team-focused facilitation, as well as staff-focused training, feedback, consultation, and incentivization.
- Total: Total of all reporting groups
Arm/Group | Facilitation, Training, Feedback, and Consultation (FTFC) Staff | Facilitation, Training, Feedback, and Consultation (FTFC) Clients | Facilitation, Training, Feedback, Consultation, and Incentivization (FTFCI) Staff | Facilitation, Training, Feedback, Consultation, and Incentivization (FTFCI) Clients | Total
Number analyzed (Participants) | 44 | 117 | 43 | 224 | 428
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 44 | 109 | 40 | 206 | 399
  >=65 years | 0 | 8 | 3 | 18 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 20 | 27 | 74 | 152
  Male | 13 | 97 | 16 | 150 | 276
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 38 | 10 | 53 | 118
  Not Hispanic or Latino | 27 | 79 | 33 | 171 | 310
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 0 | 8 | 12
  Asian | 1 | 1 | 2 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 4 | 0 | 6 | 11
  Black or African American | 11 | 51 | 21 | 129 | 212
  White | 23 | 51 | 16 | 73 | 163
  More than one race | 1 | 3 | 0 | 3 | 7
  Unknown or Not Reported | 6 | 4 | 4 | 2 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44 | 117 | 43 | 224 | 428

OUTCOME MEASURES:

1. Primary Outcome: Staff-level Implementation Consistency
Description: The cumulative number of brief interventions that each HSO staff participant implemented with HSO client participants during the implementation phase.
Time Frame: Assessed at the end of month 12
Measure: Mean (Standard Deviation); unit: client participants
Arm/Group | Facilitation, Training, Feedback, and Consultation (FTFC) Staff | Facilitation, Training, Feedback, Consultation, and Incentivization (FTFCI) Staff
Number analyzed (Participants) | 44 | 43
client participants | .73 (1.55) | 2.35 (6.67)

2. Primary Outcome: Staff-level Implementation Quality
Description: The cumulative sum quality score that each HSO staff participant demonstrated during the implementation phase. Each motivational interviewing brief intervention (MIBI) is rated on a scale from 0 (zero quality) to 12 (highest quality possible). Each individual MIBI quality score is summed to create a cumulative sum quality score. Higher scores indicated higher quality (i.e. motivational interviewing fidelity). The lower limit is zero. There is not an upper limit.
Time Frame: Assessed at the end of month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Training, Feedback, Consultation, and Facilitation: A multilevel implementation strategy
  The facilitation, training, feedback, and consultation (FTFC) Strategy: A multilevel implementation strategy that includes team-focused facilitation, as well as staff-focused training, feedback, and consultation
- Training, Feedback, Consultation, Facilitation, and P4P: An enhanced version of the multilevel implementation strategy
  The facilitation, training, feedback, consultation, and pay-for-performance (FTFC+PFP) Strategy: A multilevel implementation strategy that includes team-focused facilitation, as well as staff-focused training, feedback, consultation, and pay-for-performance.
Arm/Group | Training, Feedback, Consultation, and Facilitation | Training, Feedback, Consultation, Facilitation, and P4P
Number analyzed (Participants) | 44 | 43
score on a scale | 4.61 (9.87) | 12.39 (20.57)

3. Secondary Outcome: Staff-level Average Change (Follow-up Minus Baseline) in Their Client Participant's Days Using Primary Substance
Description: A staff-level measure representing the average level of client participant change (follow-up minus baseline) in the number of days clients used their primary substance (i.e., the substance the client identified a willingness to talk about during the MIBI) during the past 28 day
Time Frame: Assessed at 4-weeks from the baseline assessment
Measure: Mean (Standard Deviation); unit: days of reduced use
Arm/Group | Training, Feedback, Consultation, and Facilitation | Training, Feedback, Consultation, Facilitation, and P4P
Number analyzed (Participants) | 44 | 43
days of reduced use | -1.11 (4.93) | -5.95 (17.25)

4. Secondary Outcome: Staff-level Average Change (Follow-up Minus Baseline) in Their Client Participant's Generalized Anxiety Disorder 7-item (GAD-7) Score
Description: A staff-level measure of the average change (follow-up minus baseline) in their client participant's Generalized Anxiety Disorder 7-item (GAD-7) scale score. The GAD-7 ranges from 0 to 21, with higher scores indicating greater generalized anxiety. For change in the GAD-7 between baseline and follow-up (follow-up minus baseline), scores range from -20 to 20 and negative numbers are better as they indicate decreasing generalized anxiety. For this study, we examined the average GAD-7 change score that the HSO staff had with their client participants.
Time Frame: Assessed at 4-weeks from the baseline assessment
Measure: Mean (Standard Deviation); unit: change in scale score
Arm/Group | Training, Feedback, Consultation, and Facilitation | Training, Feedback, Consultation, Facilitation, and P4P
Number analyzed (Participants) | 44 | 43
change in scale score | -0.14 (3.63) | -2.63 (8.67)

ADVERSE EVENTS:
Time Frame: 1 year
Description: As also noted in the participant flow section, the Training, Feedback, Consultation, and Facilitation condition includes 161 participants, which is composed of 44 HSO staff and 117 HSO clients, whereas the Training, Feedback, Consultation, Facilitation, and Incentivization condition includes 43 HSO staff and 224 HSO clients.
Groups:
- Facilitation, Training, Feedback, and Consultation (FTFC) Clients: A multilevel implementation strategy
  The facilitation, training, feedback, and consultation (FTFC) Strategy: A multilevel implementation strategy that includes team-focused facilitation, as well as staff-focused training, feedback, and consultation
- Facilitation, Training, Feedback, Consultation, and Incentivization (FTFCI) Staff; Facilitation, Training, Feedback, Consultation, and Incentivization (FTFCI) Clients: An enhanced version of the multilevel implementation strategy
  The facilitation, training, feedback, consultation, and incentivization (FTFC + Incentivization) Strategy: A multilevel implementation strategy that includes team-focused facilitation, as well as staff-focused training, feedback, consultation, and incentivization.
Arm/Group | Facilitation, Training, Feedback, and Consultation (FTFC) Staff | Facilitation, Training, Feedback, and Consultation (FTFC) Clients | Facilitation, Training, Feedback, Consultation, and Incentivization (FTFCI) Staff | Facilitation, Training, Feedback, Consultation, and Incentivization (FTFCI) Clients
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/117 | 0/43 | 0/224
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/117 | 0/43 | 0/224
Other Adverse Events (participants affected / at risk) | 0/44 | 0/117 | 0/43 | 0/224

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/17/NCT04687917/Prot_SAP_000.pdf